CLINICAL TRIAL: NCT00005816
Title: Active Immunotherapy of Metastatic Renal Cell Carcinoma Using Autologous Dendritic Cells Transfected With Autologous Total Tumor RNA
Brief Title: Vaccine Therapy in Treating Patients With Stage III or Stage IV Kidney Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 1716; DUMC-1862-99-10; DUMC-DORIS-99124; DUMC-GCRC-839; NCI-G00-1787; CDR0000067820 (Other: NCI); 1R01CA089102-01 (NIH)
Record Dates: First submitted 2000-06-02; First posted 2004-03-23 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2008-12

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

INTERVENTIONS:
Biological: therapeutic autologous dendritic cells
Procedure: conventional surgery

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy in treating patients who have stage III or stage IV kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of autologous dendritic cells transfected with autologous total tumor RNA in patients with stage III or IV renal cell carcinoma. II. Assess the toxicity and feasibility of this treatment regimen in these patients. III. Evaluate this regimen in terms of cellular immune response, clinical response, and overall survival in these patients.

OUTLINE: This is a dose-escalation study. Patients undergo nephrectomy for tumor RNA extraction followed by leukapheresis to collect peripheral blood mononuclear cells for dendritic cell (DC) production. Patients receive autologous DC transfected with autologous renal cell carcinoma RNA both IV and intradermally on weeks 0, 2, and 4. Cohorts of 3-6 patients receive escalating doses of DC IV until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Patients are followed every 3 months for 1 year and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 18 patients will be accrued for this study over 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage III or IV renal cell carcinoma scheduled for resection of primary renal tumor No CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: At least 6 months Hematopoietic: WBC at least 3,000/mm3 Hemoglobin at least 9 mg/dL (transfusion independent) Platelet count at least 100,000/mm3 No history of bleeding disorder or other blood dyscrasias Hepatic: Bilirubin less than 2.0 mg/dL PT less than 1.5 times control No serious hepatic disease Renal: Creatinine no greater than 2.5 mg/dL Calcium less than 12 mg/dL No symptomatic hypercalcemia Cardiovascular: No serious cardiac disease (e.g., New York Heart Association class III or IV heart disease) No deep vein thrombosis Pulmonary: No serious pulmonary disease (e.g., asthma or chronic obstructive pulmonary disease) No pulmonary embolism Other: No serious chronic or acute illness that would preclude study No autoimmune disease (e.g., inflammatory bowel disease, systemic lupus erythematosus, rheumatoid arthritis, ankylosing spondylitis, scleroderma, or multiple sclerosis) No psychological impediment that would preclude study No prior malignancy within past 5 years except basal cell carcinoma, carcinoma in situ of the cervix, nonmelanomatous skin cancer, controlled superficial bladder cancer, or surgically or radiologically treated prostatic adenocarcinoma with no evidence of rising PSA for at least 12 months after treatment No active acute or chronic infection (e.g., symptomatic urinary tract infection, surgical site infection, or viral hepatitis) HIV negative Must have adequate peripheral vein access Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 6 weeks since prior immunotherapy (e.g., interleukin-2, interferon alfa, or autolymphocyte therapy) No other concurrent immunotherapy Chemotherapy: At least 6 weeks since prior chemotherapy and recovered No concurrent chemotherapy Endocrine therapy: At least 6 weeks since prior steroid therapy and recovered No concurrent steroid therapy Radiotherapy: At least 6 weeks since prior radiotherapy and recovered No concurrent local or palliative radiotherapy Surgery: See Disease Characteristics At least 6 weeks since other prior major surgery and recovered No prior radical nephrectomy Other: No concurrent immunosuppressive agents (e.g., azathioprine or cyclosporine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2000-02; Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Vieweg, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Su Z, Dannull J, Heiser A, Yancey D, Pruitt S, Madden J, Coleman D, Niedzwiecki D, Gilboa E, Vieweg J. Immunological and clinical responses in metastatic renal cancer patients vaccinated with tumor RNA-transfected dendritic cells. Cancer Res. 2003 May 1;63(9):2127-33. PMID 12727829